CLINICAL TRIAL: NCT01454063
Title: A Phase 3 Randomized, Double-Masked, Placebo-Controlled Study of the Effect of OMS302 on Intraoperative Pupil Diameter and Early Postoperative Pain in Subjects Undergoing Intraocular Lens Replacement With Phacoemulsification
Brief Title: Safety and Efficacy of OMS302 in Subjects Undergoing Intraocular Lens Replacement With Phacoemulsification
Acronym: OMS302-ILR-003
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OMS302 ILR 003
Record Dates: First submitted 2011-10-13; First posted 2011-10-18 (Estimated); Results first posted 2014-08-21 (Estimated); Last update posted 2014-08-21 (Estimated); Status verified 2014-08

CONDITIONS: Intraocular Lens Replacement
Keywords: cataract; lens replacement
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- OMS302 (Experimental): OMS302 diluted in Balanced Salt Solution and administered as irrigation solution during Intraocular Lens Replacement surgery.
  Interventions: Drug: OMS302
- Placebo (Placebo Comparator): Placebo diluted in Balanced Salt Solution and administered as irrigation solution during Intraocular Lens Replacement surgery.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OMS302 — OMS302 drug product will be supplied as a sterile, clear colorless liquid, free from particulates of foreign matter. Each vial contains a nominal 4.5 mL solution containing 60.75 millimolar (mM) phenylephrine hydrochloride (HCl) and 11.25 mM ketorolac tromethamine formulated in a 20 mM sodium citrate buffer (pH 6.3 +/- 0.5). For administration to patients, 4.4 mL of the drug product is added to a 500 mL bottle of commercially available balanced salt solution (BSS) through a syringe filter. This will achieve 4.0 mL of the drug product in a 500 mL bottle of BSS.
  Arms: OMS302
Drug: Placebo — Placebo drug product will be supplied as a sterile, clear colorless liquid, free from particulates of foreign matter. Each vial contains a nominal 4.5 mL solution containing 20 mM sodium citrate buffer (pH 6.3 +/- 0.5). For administration to patients, 4.4 mL of the drug product is added to a 500 mL bottle of commercially available BSS through a syringe filter. This will achieve 4.0 mL of the drug product in a 500 mL bottle of BSS.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety and efficacy of OMS302 (the study drug) for maintaining intraoperative mydriasis in individuals undergoing Intraocular Lens Replacement (ILR) surgery.

ELIGIBILITY:
Inclusion Criteria:

* Competent and willing to voluntarily provide informed consent
* 18 years of age or older
* In good general health needing to undergo cataract extraction or lens extraction with lens replacement surgery in one eye, under topical anesthesia

Exclusion Criteria:

* No allergies to the medications and/or the active ingredients of any of the study medications
* No medications with the same activities of the active ingredients in OMS302 for defined time intervals prior to and after surgery
* No other significant eye injuries, eye conditions or general medical conditions likely to interfere with the evaluation of the study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2011-09; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Whitaker, MD, Study Director — Omeros Corporation
Locations (16):
- United States (16):
  - Chandler, Arizona
  - Glendale, Arizona
  - Los Angeles, California
  - Cape Coral, Florida
  - Fort Myers, Florida
  - Stuart, Florida
  - Bloomington, Minnesota
  - St Louis, Missouri
  - Washington, Missouri
  - Albuquerque, New Mexico
  - New York, New York
  - Goodlettsville, Tennessee
  - Austin, Texas
  - Houston, Texas
  - San Antonio, Texas
  - Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Groups:
- OMS302: OMS302 diluted in Balanced Salt Solution (BSS) and administered as irrigation solution during Intraocular Lens Replacement surgery.
  OMS302: OMS302 drug product will be supplied as a sterile, clear colorless liquid, free from particulates of foreign matter. Each vial contains a nominal 4.5 mL of solution containing 60.75 millimolar (mM) phenylephrine hydrochloride (HCl) and 11.25 mM ketorolac tromethamine formulated in a 20 mM sodium citrate buffer (pH 6.3 +/- 0.5). For administration to patients, 4.4 mL of the drug product are added to a 500-mL bottle of commercially available BSS solution through a syringe filter, resulting in 4.0 mL of the drug product in the 500-mL bottle.
- Placebo: Placebo diluted in Balanced Salt Solution (BSS) and administered as irrigation solution during Intraocular Lens Replacement surgery.
  Placebo: Placebo drug product will be supplied as a sterile, clear colorless liquid, free from particulates of foreign matter. Each vial contains a nominal 4.5 mL of solution containing 20 mM sodium citrate buffer (pH 6.3 +/- 0.5). For administration to patients, 4.4 mL of the drug product are added to a 500-mL bottle of commercially available BSS solution through a syringe filter, resulting in 4.0 mL of the drug product in the 500-mL bottle.
Period: Randomized
Arm/Group | OMS302 | Placebo
Started | 202 | 203
Completed | 201 | 201
Not Completed | 1 | 2
Not completed — Adverse Event | 1 | 1
Not completed — Protocol Violation | 0 | 1
Period: Treated
Arm/Group | OMS302 | Placebo
Started | 201 | 201
Completed | 199 | 201
Not Completed | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- OMS302: OMS302 diluted in Balanced Salt Solution and administered as irrigation solution during Intraocular Lens Replacement surgery.
  OMS302: OMS302 drug product will be supplied as a sterile, clear colorless liquid, free from particulates of foreign matter. Each vial contains a nominal 4.5 mL of solution containing 60.75 mM phenylephrine hydrochloride (HCl) and 11.25 mM ketorolac tromethamine formulated in a 20 mM sodium citrate buffer (pH 6.3 +/- 0.5). For administration to patients, 4.4 mL of the drug product are added to a 500-mL bottle of commercially available BSS solution through a syringe filter, resulting in 4.0 mL of the drug product in the 500-mL bottle.
- Placebo: Placebo diluted in Balanced Salt Solution and administered as irrigation solution during Intraocular Lens Replacement surgery.
  Placebo: Placebo drug product will be supplied as a sterile, clear colorless liquid, free from particulates of foreign matter. Each vial contains a nominal 4.5 mL of solution containing 20 mM sodium citrate buffer (pH 6.3 +/- 0.5). For administration to patients, 4.4 mL of the drug product are added to a 500-mL bottle of commercially available BSS solution through a syringe filter, resulting in 4.0 mL of the drug product in the 500-mL bottle.
- Total: Total of all reporting groups
Arm/Group | OMS302 | Placebo | Total
Number analyzed (Participants) | 201 | 201 | 402
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (9.6) | 68.5 (9.9) | 68.4 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 119 | 111 | 230
  Male | 82 | 90 | 172

OUTCOME MEASURES:

1. Primary Outcome: Mean Area-under-the-Curve (AUC) Analysis of Change From Baseline in Pupil Diameter (mm) During Surgery
Description: Change in pupil diameter over time from surgical baseline (immediately prior to surgical incision) to the end of the surgical procedure (wound closure) was summarized using descriptive statistics by treatment arm and time-point (every minute).
  The primary analysis of the change in pupil diameter was based on the mean area-under-the-curve (AUC) pupil diameter change from baseline. First, the AUC of the pupil diameter from surgical baseline to wound closure was calculated using the trapezoidal rule. Second, the mean AUC was obtained by dividing the AUC by the total time of surgery. Third, the mean AUC of change from baseline was calculated by subtracting the baseline pupil diameter from the mean AUC.
Time Frame: from surgery baseline (pre-incision) through surgery end (time of cortical clean-up/wound closure)
Population: Subjects with interpretable video images obtained during intraocular lens replacement (ILR) procedure.
Measure: Mean (Standard Deviation); unit: mm
Groups:
- OMS302: OMS302 diluted in Balanced Salt Solution and administered as irrigation solution during Intraocular Lens Replacement surgery.
  OMS302: OMS302 drug product will be supplied as a sterile, clear colorless liquid, free from particulates of foreign matter. Each vial contains a nominal 4.5 mL of solution containing 60.75 mM phenylephrine HCl and 11.25 mM ketorolac tromethamine formulated in a 20 mM sodium citrate buffer (pH 6.3 +/- 0.5). For administration to patients, 4.4 mL of the drug product are added to a 500-mL bottle of commercially available BSS solution through a syringe filter, resulting in 4.0 mL of the drug product in the 500-mL bottle.
Arm/Group | OMS302 | Placebo
Number analyzed (Participants) | 184 | 180
mm | 0.1 (0.41) | -0.5 (0.58)
Statistical Analysis 1: Comparison: OMS302 vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — p-value based on the generalized Cochran-Mantel-Haenszel (CMH) test stratified by randomization strata; CMH-weighted mean difference (OMS - Placebo) adjusted for randomization strata; Mean Difference (Final Values) = 0.577, 95% CI [0.475 to 0.678], Standard Error of Mean 0.052

2. Secondary Outcome: Mean Area-under-the-Curve Analysis of Ocular Pain Visual Analog Scale (VAS) Score Within 12 Hours Postoperatively
Description: The primary analysis of the ocular pain VAS (where 0 = no pain and 100 = worst possible pain) was based on the mean area-under-the-curve (AUC). The AUC of the ocular pain VAS during 12 hours postoperatively was calculated by the trapezoidal rule in which the hour 11 was used to represent the time-point 10-12 hours. The mean AUC was defined as the AUC divided by the number of hours with ocular pain VAS results during the first 12 hours postoperatively.
Time Frame: 12 hours
Population: Subjects with scores at time points.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMS302 | Placebo
Number analyzed (Participants) | 201 | 201
units on a scale | 4.1 (8.07) | 9.2 (12.9)
Statistical Analysis 1: Comparison: OMS302 vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — p-value based on the generalized CMH test stratified by randomization strata; CMH-weighted mean difference (OMS302-placebo) adjusted for randomization strata; Mean Difference (Net) = -5.199, 95% CI [-7.307 to -3.091], Standard Error of Mean 1.076

3. Secondary Outcome: Photophobia at 6 Hours After Surgery (Ocular Pain and Symptoms Numerical Ordinal Scale [Numerical Rating System - NRS] Scores)
Description: Photophobia outcomes based on Ocular Pain and Symptoms Numerical Ordinal Scale (Numerical Rating System - NRS) at 6 hours postoperatively.
Time Frame: Six hours postoperatively
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | OMS302 | Placebo
Number analyzed (Participants) | 198 | 200
participants
  None | 108 | 133
  Mild | 70 | 46
  Moderate | 17 | 19
  Severe | 3 | 2
Statistical Analysis 1: Comparison: OMS302 vs Placebo; Test type: Superiority or Other; p = 0.0514, Cochran-Mantel-Haenszel — Treatment comparisons based on CMH test adjusting for randomization strata

4. Secondary Outcome: Photophobia at Day 1 After Surgery (Ocular Pain and Symptoms Numerical Ordinal Scale [Numerical Rating System - NRS] Scores)
Description: Photophobia outcomes based on Ocular Pain and Symptoms Numerical Ordinal Scale (Numerical Rating System - NRS) at Day 1 postoperatively
Time Frame: One day
Population: Subjects with scores at time point.
Measure: Number; unit: participants
Arm/Group | OMS302 | Placebo
Number analyzed (Participants) | 200 | 200
participants
  None | 125 | 90
  Mild | 48 | 63
  Moderate | 20 | 38
  Severe | 7 | 9
Statistical Analysis 1: Comparison: OMS302 vs Placebo; Test type: Superiority or Other; p = 0.0034, Cochran-Mantel-Haenszel — Treatment comparisons based on CMH test adjusting for the randomization strata

5. Secondary Outcome: Best Corrected Visual Acuity (BVCA) Log Score on Day 1
Description: Best-Corrected Visual Acuity (BCVA) summarized by the Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity log score. For subjects without a score due to inability to read the ETDRS chart, the log score was imputed as 1.6 for the purpose of treatment comparisons. Subjects without a score because the manifest refraction was not completed were excluded from the analysis.
Time Frame: One day
Population: Subject who could read well enough to obtain visual acuity score.
Measure: Mean (Standard Deviation); unit: Log score
Arm/Group | OMS302 | Placebo
Number analyzed (Participants) | 200 | 201
Log score | 0.1 (0.18) | 0.1 (0.19)
Statistical Analysis 1: Comparison: OMS302 vs Placebo; Test type: Superiority or Other; p = 0.0963, Wilcoxon rank-sum test — Treatment comparisons based on Wilcoxon rank-sum test stratified by randomization strata. For subjects without a score due to inability to read the ETDRS chart, the log score will be imputed as 1.6 for the purpose of treatment comparisons

6. Secondary Outcome: Ocular Inflammation in Summed Ocular Inflammation Score (SOIS) Grade on Day 1
Description: The mean SOIS summarized by treatment arm and time point on Day 1 postoperatively. Ocular inflammation was evaluated by measuring the anterior chamber cell count and flare using a slit lamp biomicroscope. SOIS was calculated by adding the average of subject's anterior chamber cells and flare grades. The minimum SOIS was 0 (indicating absence of inflammation), whereas the maximum SOIS was 8.
  Grading was as follows:
  Anterior Chamber Cells: Grade None = 0/no cells; Grade Mild = +1/1-5 cells; Grade Moderate = +2/6-15 cells; Grade Severe = +3/16-30 cells; Grade Very Severe = +4/>30 cells.
  Anterior Chamber Flare: Grade None = 0/no Tyndall effect; Grade Mild = +1/barely discernable Tyndall effect; Grade Moderate = +2/moderately intense Tyndall beam in anterior chamber; Grade Severe = +3/severely intense Tyndall beam; Grade Very Severe = +4/very severely intense Tyndall beam with a white and milky appearance to the aqueous
Time Frame: One day
Population: Subjects with score at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMS302 | Placebo
Number analyzed (Participants) | 201 | 201
units on a scale | 2.7 (1.1) | 2.9 (1.4)
Statistical Analysis 1: Comparison: OMS302 vs Placebo; Test type: Superiority or Other; p = 0.0532, Cochran-Mantel-Haenszel — Treatment comparisons are based on generalized CMH test stratified by randomization strata

7. Secondary Outcome: Ocular Pain VAS Score After Day of Surgery - Day 1
Description: Pain VAS scores (where 0 = no pain and 100 = worst possible pain) after the day of surgery summarized by treatment arm and time-point.
Time Frame: One day
Population: Number of subjects with scores at time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | OMS302 | Placebo
Number analyzed (Participants) | 201 | 201
units on a scale | 5.9 (13.3) | 14.2 (21.4)
Statistical Analysis 1: Comparison: OMS302 vs Placebo; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Generalized CMH test stratified by randomization strata

ADVERSE EVENTS:
Time Frame: 14 days post-surgery.
Arm/Group | OMS302 | Placebo
Serious Adverse Events (participants affected / at risk) | 1/201 | 0/201
Other Adverse Events (participants affected / at risk) | 156/201 | 154/201
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OMS302 (N=201) | Placebo (N=201)
electrocution (General disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OMS302 (N=201) | Placebo (N=201)
eye pain (Eye disorders) | 88 | 86
eye inflammation (Eye disorders) | 60 | 58
anterior chamber inflammation (Eye disorders) | 19 | 21
headache (Nervous system disorders) | 5 | 14
intraocular pressure increased (Investigations) | 7 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI agreed not to publish or otherwise to disclose Study data without prior written consent from the sponsor for a period of 24 months following Study completion or until data are published in a combined publication (whichever occurs first). The sponsor can review communications containing results prior to public release and embargo those communications for a period that is no longer than 60 days from the date of receipt of the non-public communication. The sponsor cannot extend the embargo.